CLINICAL TRIAL: NCT00162682
Title: A Phase III, Randomized, Non-inferiority Trial Comparing the Standard Viral Load Based Antiretroviral Monitoring Strategy With a CD4 Based Monitoring Strategy Among Antiretroviral Naive Immunocompromised Adults in Thailand
Brief Title: Monitoring Highly Active Antiretroviral Therapy in HIV-infected Parents in Thailand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Marc Lallemant, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD042964 (NIH); NCT00197626 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-13 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections
Keywords: HIV; Highly Active Antiretroviral Therapy; Monitoring; Viral load; CD4; Thailand; Future Drug Options; Resistance; Developing Country; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): * VL-S, the standard viral load (VL) based monitoring strategy, where switching is performed when VL is confirmed (within one month) above 400 copies per mL.
  Interventions: Procedure: Antiretroviral Drug Combination Switching Criteria
- 2 (Experimental): CD4-S, the alternative CD4 based monitoring strategy where switching is performed when a confirmed (within one month) relative decline in CD4 count of more than 30% from peak values is observed within 200 cells from baseline.
  Interventions: Procedure: Antiretroviral Drug Combination Switching Criteria

INTERVENTIONS:
Procedure: Antiretroviral Drug Combination Switching Criteria — Antiretroviral treatment will use the standard viral load (VL) based monitoring strategy, where switching is performed when VL is confirmed (within one month) above 400 copies per mL.
  Arms: 1
Procedure: Antiretroviral Drug Combination Switching Criteria — Antiretroviral treatment is monitored using a CD4 based monitoring strategy where switching is performed when a confirmed (within one month) relative decline in CD4 count of more than 30% from peak values is observed within 200 cells from baseline.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if a decision to switch to a subsequent antiretroviral regimen based upon the CD4 cell count rather than the standard switching strategy based on viral load could ensure the same immunological and clinical outcome and preserve future treatment options in AIDS patients

DETAILED DESCRIPTION:
Implementation of highly active antiretroviral therapy (HAART) has led to a substantial decrease in HIV-related mortality and morbidity. Current guidelines emphasize maximal and durable viral load suppression. However, while the goal of therapy is the restoration of immunity, treatment failure is usually defined as the inability to maintain undetectable viral load, without regard to immune function. This situation often leads to a rapid sequence of therapeutic switches, thus narrowing therapeutic options over time. A monitoring strategy driven primarily by the patient's immune restoration would most likely be as effective in preventing disease progression, would lead to fewer changes in HAART regimens and would be considerably simpler and cost effective.

Subjects will be randomly assigned to one of two switching strategies:

* VL-S, the standard viral load (VL) based monitoring strategy, where switching is performed when VL is confirmed (within one month) above 400 copies per mL.
* CD4-S, the alternative CD4 based monitoring strategy where switching is performed when a confirmed (within one month) relative decline in CD4 count of more than 30% from peak values is observed within 200 cells from baseline.

The initial HAART regimen will be a NNRTI+NRTI containing regimen and the second line regimen will be a PI containing regimen, subsequent regimens will be chosen individually based on tolerance, previous drugs used, resistance profile, and drugs available. Patients will be followed until the end of the study (maximum of 5 years for the first enrollee, three years for the last enrollee).

ELIGIBILITY:
Eligibility Criteria:

Patients fulfilling the following criteria are eligible:

* At least 18 years of age
* Confirmed HIV infection: two positive serology results from two different blood draws are required for documentation of HIV infection.
* Antiretroviral drug naïve with the exception of short course of antiretrovirals received in the context of the prevention of mother to child HIV transmission
* Need for antiretroviral treatment
* Willingness to receive a long-term treatment for the HIV infection, according to the study schedule at the participating site
* Signed informed consent to participate in the study (the patient's legal guardian may give his/her consent if the patient cannot provide consent)
* Does not present an exclusion criteria to the knowledge of the site investigator

Inclusion Criteria:

Eligible patients fulfilling the following criteria can be enrolled in the study:

* Meeting all eligibility criteria
* Two CD4+ cell counts between 50 and 250 cells/mm3 performed within the last six months before enrolment (CD4 cell count should be assessed at least 2 weeks apart from any acute infection)
* Willingness to modify antiretroviral therapy in accordance with the randomized switching scheme assignment
* Subject understands that study drugs will be supplied for free by the study only during participation in the study. After discontinuation of the study, patients will be taken care of in the National ARV Access Program.

Exclusion Criteria:

* For women, pregnancy
* For women of child bearing potential, lack of willingness to follow an effective method of contraception (in case, during the study, a woman wants to become pregnant or becomes pregnant, she should inform the physician immediately for best therapeutic decision)
* Chronic hepatitis B or C
* Acute hepatitis within 30 days of study entry.
* Acute HIV infection, as it can be established with the date of last negative serology less than one year before enrollment and the history of the patient disease
* Co-enrollment in another study without prior written agreement of the study team
* Psycho-social environment or condition which, in the physician's opinion, makes adherence to the protocol highly unlikely.
* Pre-existing diabetes mellitus (prior gestational diabetes is allowed).
* The following laboratory values: hemoglobin < 8.0 mg/dl, absolute neutrophil count < 1000 cells/mm3, ALT, AST or total bilirubin value > 5.0 x ULN, serum creatinine > 1.0 x ULN, platelet count < 50,000/mm3, pancreatic amylase >2.0 x ULN or lipase > 2.0 X ULN, or total amylase > 2.0 X ULN plus symptoms of pancreatitis.
* Severe illness, grade 3 or 4 laboratory exam values not resolved within one month of enrollment without previous agreement of the PHPT attending physician
* Any clinically significant condition (other than HIV infection) which, in the investigator's opinion, would interfere with the conduct of the study.
* Current active substance or alcohol abuse that would interfere with participation in the study.
* Condition(s) that contraindicate all the first line regimens proposed in this study.
* Chemotherapy for active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2005-05; Primary Completion 2010-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Proportion of "clinical failures" defined as confirmed CD4 count below 50/mm3, first or new AIDS-defining event, or death | After 3 years of follow-up

SECONDARY OUTCOMES:
The number of therapeutic options left taking into account drugs exhausted cross-resistance mutations and shared toxicities | After 3 years of follow-up
The secondary endpoint related to safety will be time to the first development of grade 3 or grade 4 sign, symptom, and laboratory abnormality. | During 3 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, MD, Principal Investigator — Institut de Recherche pour le Developpement & Harvard School of Public Health
Locations (20):
- Thailand (20):
  - Buddhachinaraj Hospital, Bangkok, Bangkok
  - Chacheongsao Hospital, Chacheongsao, Chacheongsao
  - Prapokklao Hospital, Prapokklao, Muang, Changwat Chanthaburi
  - Mae Chan Hospital, Mae Chan, Changwat Chiang Rai
  - Chonburi Hospital, Muang, Chonburi, Changwat Chon Buri
  - Regional Health Promotion Centre 6,, Khon Kaen, Changwat Khon Kaen
  - Lampang Hospital, Lampang, Changwat Lampang
  - Lamphun Hospital, Muang, Changwat Lamphun
  - Nong Khai Hospital, Muang, Nong Khai, Changwat Nong Khai
  - Phayao Provincial Hospital, Muang, Changwat Phayao
  - Ratchaburi Hospital, Muang, Ratchaburi, Changwat Ratchaburi
  - Rayong Hospital, Rayong, Changwat Rayong
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - Sanpatong Hospital, Sanpatong, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Muang, Chiangrai, Chiangrai
  - Mahasarakam Hospital, Muang, Mahasarakam
  - Maharaj Nakornratchasrima Hospital, Muang, Nakornratchasrima, Nakornratchasrima
  - Samutprakarn Hospital, Samutprakarn, Samutprakarn
  - Samutsakorn Hospital, Muang, Samutsakorn, Samutsakorn

REFERENCES:
- [Result] Jourdain G, Ngo-Giang-Huong Nicole, Le Coeur S, Traisaithit P, Barbier S, Techapornroong M, Banchongkit S, Buranabanjasatean S, Halue G, Lallemant M, and The PHPT-3 study group. PHPT-3: A Randomized Clinical Trial Comparing CD4 versus Viral Load (VL) Antiretroviral Therapy Monitoring/Switching Strategies in Thailand. 18th Conference on Retroviruses and Opportunistic Infections, 27 February-2 March, 2011,Boston, USA. Oral Presentation #44.
- [Result] Cressey TR, Urien S, Hirt D, Halue G, Techapornroong M, Bowonwatanuwong C, Leenasirimakul P, Treluyer JM, Jourdain G, Lallemant M; PHPT-3 Team. Influence of body weight on achieving indinavir concentrations within its therapeutic window in HIV-infected Thai patients receiving indinavir boosted with ritonavir. Ther Drug Monit. 2011 Feb;33(1):25-31. doi: 10.1097/FTD.0b013e3182057f6f. PMID 21233689
- [Derived] Jourdain G, Le Coeur S, Ngo-Giang-Huong N, Traisathit P, Cressey TR, Fregonese F, Leurent B, Collins IJ, Techapornroong M, Banchongkit S, Buranabanjasatean S, Halue G, Nilmanat A, Luekamlung N, Klinbuayaem V, Chutanunta A, Kantipong P, Bowonwatanuwong C, Lertkoonalak R, Leenasirimakul P, Tansuphasawasdikul S, Sang-A-Gad P, Pathipvanich P, Thongbuaban S, Wittayapraparat P, Eiamsirikit N, Buranawanitchakorn Y, Yutthakasemsunt N, Winiyakul N, Decker L, Barbier S, Koetsawang S, Sirirungsi W, McIntosh K, Thanprasertsuk S, Lallemant M; PHPT-3 study team. Switching HIV treatment in adults based on CD4 count versus viral load monitoring: a randomized, non-inferiority trial in Thailand. PLoS Med. 2013 Aug;10(8):e1001494. doi: 10.1371/journal.pmed.1001494. Epub 2013 Aug 6. PMID 23940461
- See also: Related Info — http://www.phpt.org